CLINICAL TRIAL: NCT01410110
Title: Cognitive Remediation and Work Therapy in the Initial Phase of Substance Abuse Treatment
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Yale University (Other)
Responsible Party: Principal Investigator, Morris D. Bell, Professor, Yale University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1011007601; R21DA030744-02 (NIH)
Record Dates: First submitted 2011-08-02; First posted 2011-08-04 (Estimated); Results first posted 2015-01-19 (Estimated); Last update posted 2015-01-19 (Estimated); Status verified 2014-12

CONDITIONS: Substance Abuse; Substance Dependence; Cognitive Impairment
Keywords: Substance Abuse; Substance Dependence; Cognitive Impairment
MeSH Terms: conditions — Substance-Related Disorders; Cognitive Dysfunction | interventions — Cognitive Training

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cognitive Training + Work Therapy (Experimental): Cognitive Training using auditory and visual Positscience software 5 hours/per week for 13 weeks.
  Work Therapy for 15 hours per week at half minimum wage doing entry level duties at medical center job sites, supervised by regular medical center staff.
  Interventions: Behavioral: Cognitive Training + Work Therapy
- Work Therapy Only (Active Comparator): Same work therapy but for 20 hours per week.
  Interventions: Behavioral: Work Therapy

INTERVENTIONS:
Behavioral: Cognitive Training + Work Therapy — Cognitive training for 5 hours per week for 13 weeks and 15 hours of work therapy
  Arms: Cognitive Training + Work Therapy
Behavioral: Work Therapy — 20 hours per week of work therapy
  Arms: Work Therapy Only

SUMMARY:
The initial phase of substance abuse treatment is a vulnerable period for relapse. Cognitive impairments are common during this phase and may reduce the ability to benefit from other forms of substance abuse and rehabilitation services. The study compares a rehabilitation program that combines work therapy with computer-based cognitive training of attention, memory and executive functions to work therapy alone in a 3 months outpatient substance abuse program. It is hypothesized that cognitive training will increase days of sobriety during the active intervention and better substance abuse outcomes at 6 month follow-up.

DETAILED DESCRIPTION:
This proposal aims to pilot test a cognitive remediation therapy (CRT) combined with work therapy (WT) as an adjunct to the initial phase of outpatient substance abuse treatment. There is ample research evidence of cognitive impairment across substance abuse disorders, particularly in the early phase of recovery. Cognitive impairment has been associated with poorer substance abuse treatment outcomes and may be remediated through programs of exercises that target these impairments. The investigators have previously reported on a model of providing CRT with work therapy (WT) in an outpatient context for people with psychotic disorders, which showed significant improvements in executive function and working memory, and in important functional outcomes such as work performance and sustained work activity. The investigators propose to apply this same approach to a sample of participants recruited from a 30-day residential program for substance abusers who are beginning their recovery. When they are discharged, they will be able to continue WT, which may encourage their engagement in CRT and in substance abuse outpatient services.

Our Specific Aims are: 1. Test the feasibility and tolerability of CRT & WT in the early phase of substance abuse treatment. 2. Obtain effect size for CRT & WT compared to WT alone on a primary substance abuse outcome measure (Days of Use) for a future R01 RCT submission. 3. Obtain effect sizes for secondary outcomes (e.g. neurocognition).

The investigators propose to accomplish these aims by randomizing 50 participants who wish to receive WT services into two conditions: 25 will be assigned to 15 hours of WT plus 5 hours of CRT each week (CRT+WT) and 25 will be assigned to an active control of 20 hours of WT. The active intervention will be for 13 weeks. CRT will be comprised of a repetitive training on a hierarchy of progressive visual and auditory exercise from Positscience. WT will involve paid work activity in a placement of their choosing on the medical center campus. Participants will be paid the same hourly rate (half federal minimum wage) for their time in CRT and WT. Comprehensive assessments will be performed at intake, 3 months and 6 months. These will include substance abuse, cognitive, and psychosocial outcomes as well as adherence to treatment. During the 3 months of active intervention participants will have weekly observed urine toxicology screens, breathalyzer tests and PDA assessments, as well as monthly work performance evaluations. Data analyses will include random effects regression models, as well as models of moderator and mediator effects on the primary outcome of PDA. If meaningful effects are found, these results will guide a subsequent R01 submission.

ELIGIBILITY:
Inclusion Criteria:

* In the initial phase of treatment for substance abuse or dependence at VACHS.
* Fluency in English 6th grade or higher reading level DSM-IV criteria for any current drug use disorder
* Willingness to attend follow-up assessments at 13 and 26 weeks
* Willingness to submit to observed urine toxicology and breathalyzer screenings

Exclusion Criteria:

* Untreated psychotic disorder
* Current prescribed treatment of opioids or benzodiazepines
* Having a legal case that may lead to incarceration during study period
* Residential plans that would interfere with participation
* Developmental disability or medical illness that may significantly compromise cognition or prevent work activity

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2010-12; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Morris D Bell, Ph.D., Principal Investigator — Yale University School of Medicine and VACHS
Locations (1):
- VA Connecticut Healthcare System, West Haven, Connecticut, United States

REFERENCES:
- [Derived] Bell MD, Laws HB, Petrakis IB. A randomized controlled trial of cognitive remediation and work therapy in the early phase of substance use disorder recovery for older veterans: Neurocognitive and substance use outcomes. Psychiatr Rehabil J. 2017 Mar;40(1):94-102. doi: 10.1037/prj0000211. Epub 2016 Oct 10. PMID 27732034
- [Derived] Bell MD, Vissicchio NA, Weinstein AJ. Cognitive Training and Work Therapy for the Treatment of Verbal Learning and Memory Deficits in Veterans With Alcohol Use Disorders. J Dual Diagn. 2016;12(1):83-9. doi: 10.1080/15504263.2016.1145779. PMID 26828571
- [Derived] Bell MD, Vissicchio NA, Weinstein AJ. Visual and verbal learning deficits in Veterans with alcohol and substance use disorders. Drug Alcohol Depend. 2016 Feb 1;159:61-5. doi: 10.1016/j.drugalcdep.2015.11.007. Epub 2015 Dec 2. PMID 26684868

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment was by referral from clinicians at VA Substance Abuse program including a 21 day substance abuse day program and a 30 day residential program. Recruitment began in January 2011 and was completed in March 2014.
Pre-assignment Details: Following informed consent, participants completed baseline assessments and their VA medical record was reviewed to determine whether they met inclusion/exclusion criteria.
Groups:
- Cognitive Training + Work Therapy: Cognitive Training using auditory and visual Positscience software 5 hours/per week for 13 weeks.
  Work Therapy for 15 hours per week at half minimum wage doing entry level duties at medical center job sites, supervised by regular medical center staff.
  Cognitive Training + Work Therapy: Cognitive training for 5 hours per week for 13 weeks and 15 hours of work therapy
Period: Overall Study
Arm/Group | Cognitive Training + Work Therapy | Work Therapy Only
Started | 24 | 24
Randomization | 24 | 24
3 Months (End of Intervention) | 20 | 22
6 Month Follow-up | 20 | 22
Completed | 20 | 22
Not Completed | 4 | 2
Not completed — Withdrawal by Subject | 4 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cognitive Training + Work Therapy | Work Therapy Only | Total
Number analyzed (Participants) | 24 | 24 | 48
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.3 (9.7) | 53.8 (7.4) | 52.55 (8.55)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 3
  Male | 22 | 23 | 45
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 24 | 24 | 48
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 3 | 3
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 11 | 13 | 24
  White | 13 | 7 | 20
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0
Marital Status [Number; unit: participants]
  Married | 3 | 6 | 9
  Never Married | 5 | 8 | 13
  Divorced/Widowed | 16 | 10 | 26
Axis 1 Primary Diagnosis [Number; unit: participants]
  Alcohol Use Disorder | 13 | 15 | 28
  Cocaine | 3 | 7 | 10
  Opiods | 6 | 0 | 6
  Other | 2 | 2 | 4
Education [Mean (Standard Deviation); unit: years] | 13.2 (1.6) | 12.21 (1.5) | 12.71 (1.55)
Felony Convictions [Number; unit: participants]
  Yes | 11 | 12 | 23
  No | 13 | 12 | 25
Disability (SSDI or VA Service Connected) [Number; unit: participants]
  Yes | 2 | 3 | 5
  No | 22 | 21 | 43
Global Assessment of Function (GAF) [Mean (Standard Deviation); unit: units on a scale] — The Global Assessment of Function Scale range is from 1 to 100. Higher scores indicate better functioning.
  units on a scale | 45.17 (3.6) | 47.67 (5.9) | 46.42 (4.75)

OUTCOME MEASURES:

1. Primary Outcome: Days of Sobriety in First 90 Days
Description: Abstinence will be determined by toxicology screening, breathalyzer and substance abuse calendar weekly during 3 months of active intervention. Days of sobriety has a range of 0 to 90 with higher being a better outcome.
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: Days of Sobriety
Arm/Group | Cognitive Training + Work Therapy | Work Therapy Only
Number analyzed (Participants) | 20 | 22
Days of Sobriety | 87.3 (7.8) | 84.64 (18.2)
Statistical Analysis 1: Comparison: Cognitive Training + Work Therapy vs Work Therapy Only; t-test for equality of means; Test type: Superiority or Other; p = .55, t-test, 2 sided — a prior threshold p < .05; df = 40; Mean Difference (Final Values) = -2.66, 95% CI 2-sided [-11.57 to 6.25], Standard Error of Mean 4.41

2. Secondary Outcome: Attention Index
Description: Index comprised on Trails A and Continuous Performance Test. T scores for the assessments are averaged. T scores range from 30 to 80 with a mean of 50. Higher scores are better.
Time Frame: Baseline, 3 month and 6 month follow-up
Measure: Mean (Standard Deviation); unit: T Scores
Arm/Group | Cognitive Training + Work Therapy | Work Therapy Only
Number analyzed (Participants) | 24 | 24
T Scores
  Baseline | 48.08 (8.26) | 41.79 (8.87)
  3 Month | 48.17 (8.74) | 43.19 (9.54)
  6 Month | 50.36 (10.14) | 43.55 (10.24)
Statistical Analysis 1: Comparison: Cognitive Training + Work Therapy vs Work Therapy Only; F Test (df = 1,39.32), Type III Fixed Effects for Time X Condition; Test type: Superiority or Other; p = .86, Mixed Models Analysis — Time X Condition; Mixed Models allows for all randomized participants (N=48) to be included in the model; Slope = .162, 95% CI 2-sided [-1.73 to 2.05], Standard Error of Mean .94

3. Primary Outcome: Days of Use in Prior 30 Days
Description: Days of Use based on Time-Line Follow-back, Toxicology Screen, Breathalyzer, and Chart Review. The range at 6 month follow-up is 0 to 30 days of use with more days being a worse outcome.
Time Frame: 30 Days Prior to 6 month follow-up
Measure: Mean (Standard Deviation); unit: Days of Use
Arm/Group | Cognitive Training + Work Therapy | Work Therapy Only
Number analyzed (Participants) | 20 | 22
Days of Use | 4.35 (9.44) | 1.86 (5.96)
Statistical Analysis 1: Comparison: Cognitive Training + Work Therapy vs Work Therapy Only; Test type: Superiority or Other; p < .31, t-test, 2 sided — a priori threshold p < .05; Mean Difference (Final Values) = -2.49, 95% CI 2-sided [-7.36 to 2.39], Standard Error of Mean 2.41

4. Primary Outcome: Weeks of Sobriety
Description: 0 to 26 Weeks. Higher number of Weeks is better.
Time Frame: 26 weeks
Population: 1 additional participant in Work Therapy Only had missing data for this variable.
Measure: Mean (Standard Deviation); unit: Weeks
Arm/Group | Cognitive Training + Work Therapy | Work Therapy Only
Number analyzed (Participants) | 20 | 21
Weeks | 23.80 (2.8) | 23.95 (3.25)
Statistical Analysis 1: Comparison: Cognitive Training + Work Therapy vs Work Therapy Only; Test type: Superiority or Other; p = .87, t-test, 2 sided — a priori threshold p < .05; df=39; Mean Difference (Final Values) = .152, 95% CI 2-sided [-1.77 to 2.08], Standard Error of Mean .952

5. Secondary Outcome: Processing Speed Index
Description: Wechsler Adult Intelligence Scale (WAIS) Digit Coding and Symbol Search. T scores for the assessments are averaged. T scores range from 30 to 80 with a mean of 50. Higher scores are better.
Time Frame: Baseline, 3 Months, 6 Months
Measure: Mean (Standard Deviation); unit: T Scores
Arm/Group | Cognitive Training + Work Therapy | Work Therapy Only
Number analyzed (Participants) | 24 | 24
T Scores
  Baseline | 49.42 (7.46) | 45.06 (9.14)
  3 Months | 49.61 (9.04) | 45.57 (10.03)
  6 Months | 50.42 (9.39) | 46.90 (9.54)
Statistical Analysis 1: Comparison: Cognitive Training + Work Therapy; Type III Fixed Effects for Time X Condition F Test (df = 1,36.86); Test type: Superiority or Other; p = .67, Mixed Models Analysis; Time X Condition; Slope = -.37, 95% CI 2-sided [-2.07 to 1.33], Standard Error of Mean .84

6. Secondary Outcome: Verbal and Visual Learning and Memory
Description: Brief Visual-Spatial Memory Test (BVMT) and Hopkins Verbal Learning and Memory Test (HVLT). Total Score T Scores for tests were averaged. T score range is 30 to 80 with a mean of 50. Higher scores are better.
Time Frame: Baseline, 3 Months, 6 Months
Measure: Mean (Standard Deviation); unit: T Scores
Arm/Group | Cognitive Training + Work Therapy | Work Therapy Only
Number analyzed (Participants) | 24 | 24
T Scores
  Baseline | 38.13 (9.39) | 33.5 (10.89)
  3 Months | 40.48 (8.3) | 36.67 (11.1)
  6 Months | 39.5 (11.3) | 38.3 (9.9)
Statistical Analysis 1: Comparison: Cognitive Training + Work Therapy vs Work Therapy Only; Type III Fixed Effects for Time X Condition, F Test F (df = 1,42.4); Test type: Superiority or Other; p = .50, Mixed Models Analysis; Time X Condition; Slope = -.42, 95% CI 2-sided [-1.67 to .83], Standard Error of Mean .62

7. Secondary Outcome: Verbal and Visual Working Memory
Description: WAIS Digit Span and Wechsler Memory Scale (WMS) Spatial Span. T Scores are averaged. T Scores range from 30 to 80 with a mean of 50. Higher scores are better.
Time Frame: Baseline, 3 Month, 6 Months
Measure: Mean (Standard Deviation); unit: T Scores
Arm/Group | Cognitive Training + Work Therapy | Work Therapy Only
Number analyzed (Participants) | 24 | 24
T Scores
  Baseline | 45.43 (6.26) | 43.25 (8.49)
  3 Month | 46.25 (12.1) | 40.62 (7.5)
  6 Month | 50.00 (9.37) | 42.62 (9.3)
Statistical Analysis 1: Comparison: Cognitive Training + Work Therapy vs Work Therapy Only; Type III Fixed Effects Time X Condition F Test (df = 1,70.15); Test type: Superiority or Other; p = .008, Mixed Models Analysis; Time X Condition; Slope = 1.16, 95% CI 2-sided [.32 to 2.01], Standard Error of Mean .42

8. Secondary Outcome: Executive Function
Description: Mazes, Wisconsin Card Sorting Task (WCST) Perseverative Error, Non-Perseverative Error, Conceptual Level. T Scores for each variable were averaged together. T Scores have a range of 30 to 80 with a mean of 50. Higher scores are better.
Time Frame: Baseline, 3 Months, 6 Months
Measure: Mean (Standard Deviation); unit: T Scores
Arm/Group | Cognitive Training + Work Therapy | Work Therapy Only
Number analyzed (Participants) | 24 | 24
T Scores
  Baseline | 45.11 (6.75) | 42.59 (7.72)
  3 Month | 48.8 (8.4) | 43.26 (8.7)
  6 Month | 49.53 (9.8) | 43.8 (8.3)
Statistical Analysis 1: Comparison: Cognitive Training + Work Therapy vs Work Therapy Only; Type III Fixed Effects Time X Condition F Test (df = 1,37.8); Test type: Superiority or Other; p = .03, Mixed Models Analysis; Time X Condition; Slope = 2.025, 95% CI 2-sided [.169 to 3.93], Standard Error of Mean .93

9. Secondary Outcome: Global Index
Description: Comprised of the average of 5 Index T Scores (Attention, Processing Speed, Visual and Verbal Memory and Learning, Working Memory and Executive Function). T Scores range from 30 to 80 with a mean of 50. Higher scores are better.
Time Frame: Baseline, 3 Months, 6 Months
Measure: Mean (Standard Deviation); unit: T Scores
Arm/Group | Cognitive Training + Work Therapy | Work Therapy Only
Number analyzed (Participants) | 24 | 24
T Scores
  Intake | 45.23 (5.36) | 41.25 (7.54)
  3 Months | 46.63 (7.55) | 41.86 (7.66)
  6 Months | 47.95 (7.95) | 43.05 (7.68)
Statistical Analysis 1: Comparison: Cognitive Training + Work Therapy vs Work Therapy Only; Type III Fixed Effects for Time X Condition F Test (df = 1,39.8); Test type: Superiority or Other; p = .17, Mixed Models Analysis — a priori p-value is .05. for two-tailed test. Positive estimated value is in the direction of the experimental condition; Time X Condition; Slope = 3.86, 95% CI 2-sided [-1.73 to 9.46], Standard Error of Mean 2.77

ADVERSE EVENTS:
Time Frame: Entire length of study
Arm/Group | Cognitive Training + Work Therapy | Work Therapy Only
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/24
Other Adverse Events (participants affected / at risk) | 0/24 | 0/24

LIMITATIONS AND CAVEATS:
Use of WT limited recruitment to only those willing to participate in a work program for 13 weeks, reducing generalizability. WT may have powerful effects on sobriety that obscured benefits of CRT. As a pilot, this study was not adequately powered.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No